CLINICAL TRIAL: NCT00710034
Title: Oral Tobacco as a Harm Reduction Product: Study 2 - Efficacy of Oral Tobacco Products Compared to Medicinal Nicotine for Complete Cigarette Substitution and Among Non-abstainers, for Reduction in Cigarette Smoking
Brief Title: Efficacy of Oral Tobacco Products Compared to a Medicinal Nicotine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1R01 CA135884-2; 1R01CA135884 (NIH)
Record Dates: First submitted 2008-07-02; First posted 2008-07-03 (Estimated); Results first posted 2017-12-06 (Actual); Last update posted 2017-12-06 (Actual); Status verified 2017-10

CONDITIONS: Tobacco Use Disorder
Keywords: Oral Tobacco Products; Snus; Smoking Substitution; Harm Reduction; Biomarkers of Tobacco Exposure
MeSH Terms: conditions — Tobacco Use Disorder; Harm Reduction | interventions — Tobacco, Smokeless; Nicotine Chewing Gum

STUDY DESIGN:
Masking Description: This was an open label trial.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nicotine Gum (Active Comparator): Nicotine replacement therapy (4 mg nicotine gum) was provided to the participants for an 12 weeks. Participants were encouraged to completely substitute nicotine gum for cigarettes and asked to use at least 6-8 pieces a day or optimally every 1-2 h and more if necessary. They were advised to reduce consumption by half during weeks 7-9 and three-quarters during weeks 10-12.
  Interventions: Drug: Nicotine Gum
- Snus (Experimental): Oral tobacco (Camel Snus) was provided to the participants for an 12 weeks. Participants were encouraged to completely substitute snus for cigarettes and asked to use at least 6-8 pieces a day or optimally every 1-2 h and more if necessary. They were advised to reduce consumption by half during weeks 7-9 and three-quarters during weeks 10-12.
  Interventions: Other: Oral tobacco

INTERVENTIONS:
Other: Oral tobacco — Snus
  Other Names: Camel Snus
  Arms: Snus
Drug: Nicotine Gum — 4 mg Nicotine gum
  Other Names: Nicorette
  Arms: Nicotine Gum

SUMMARY:
For the primary goals, we hypothesize that 1) the oral tobacco product will be more efficacious than the medicinal nicotine product in substituting for smoking cigarettes; 2) among non-abstainers, the oral tobacco product will lead to greater reduction in cigarette smoking than medicinal nicotine; and 3) a higher rate of oral tobacco compared to medicinal nicotine use will be observed during and beyond the treatment period.

For the secondary goals, we hypothesize that 1) both products will equally reduce withdrawal symptoms from cigarette abstinence; and 2) the toxicant exposure and toxicity will be reduced dramatically when smokers switch from cigarettes to each of these products; however, this reduction will be greater with the use of medicinal nicotine.

DETAILED DESCRIPTION:
This second study under "Oral Tobacco as a Harm Reduction Product" grant is a clinical trial. Subjects will be randomized to the brand of smokeless tobacco that is determined to be most effective in Study 1 or to nicotine gum for 12 weeks to compare complete substitution for smoking. The secondary aims are to determine the effects of the products on biomarkers of exposure and toxicity. Other secondary aim includes examining the effects of the two products on withdrawal symptoms. Two sites will be used for these studies: University of Minnesota and Oregon Research Institute (ORI).

ELIGIBILITY:
Inclusion Criteria:

* smoking at least 10 cigarettes daily for the past year,
* in good physical health (no unstable medical condition;
* no contraindications for medicinal nicotine, as appropriate for the study, stable, good mental health (e.g., no recent unstable or untreated psychiatric diagnosis, including substance abuse, as determined by the DSM-IV criteria).

Exclusion Criteria:

Subjects must not be currently using other tobacco or nicotine products; Female subjects cannot be pregnant or nursing.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 391 (Actual)
Dates: Start 2010-04; Primary Completion 2013-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dorothy Hatsukami, Ph.D., Principal Investigator — University of Minnesota
Locations (2):
- United States (2):
  - University of Minnesota, Minneapolis, Minnesota
  - Oregon Research Institute, Eugene, Oregon

IPD SHARING:
Plan to Share IPD: Yes
We will share data with both internal and external researchers. Those external researchers interested in accessing the data will be required to submit a data analyses proposal with specific aims, hypotheses, and data analyses plan. These proposals will be reviewed by the investigative team. The requested data will then be provided that includes the variable list, raw data and description of the measures and methods of data collection.

REFERENCES:
- [Background] Hatsukami DK, Severson H, Anderson A, Vogel RI, Jensen J, Broadbent B, Murphy SE, Carmella S, Hecht SS. Randomised clinical trial of snus versus medicinal nicotine among smokers interested in product switching. Tob Control. 2016 May;25(3):267-74. doi: 10.1136/tobaccocontrol-2014-052080. Epub 2015 May 19. PMID 25991608

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Cigarette smokers interested in completely switching to snus or nicotine gum were recruited from Minneapolis/St Paul, Minnesota, and Eugene, Oregon.
Groups:
- Nicotine Gum: Nicotine replacement therapy
  Nicotine Gum: 4 mg Nicotine gum
- Snus: Oral tobacco
  Oral tobacco: Snus
Period: Completed 6 Weeks of Treatment
Arm/Group | Nicotine Gum | Snus
Started | 195 | 196
Completed | 154 (Completed 6 weeks of treatment for primary outcome assessment: N=154) | 149 (Completed 6 weeks of treatment for primary outcome assessment: N=149)
Not Completed | 41 | 47
Not completed — Adverse Event | 5 | 12
Not completed — Lack of Efficacy | 12 | 8
Not completed — Lost to Follow-up | 15 | 17
Not completed — Product dissatisfaction | 2 | 6
Not completed — Withdrawal by Subject | 6 | 4
Not completed — Physician Decision | 1 | 0
Period: Completed 12 Weeks of Treatment
Arm/Group | Nicotine Gum | Snus
Started | 154 | 149
Completed | 141 | 138
Not Completed | 13 | 11
Not completed — Adverse Event | 0 | 1
Not completed — Lack of Efficacy | 0 | 2
Not completed — Lost to Follow-up | 5 | 5
Not completed — Product Dissatisfaction | 0 | 1
Not completed — Withdrawal by Subject | 8 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nicotine Gum | Snus | Total
Number analyzed (Participants) | 195 | 196 | 391
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 195 | 196 | 391
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.9 (12.5) | 43.2 (12.5) | 43.9 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 95 | 89 | 184
  Male | 100 | 107 | 207
Region of Enrollment [Number; unit: participants]
  United States | 195 | 196 | 391

OUTCOME MEASURES:

1. Primary Outcome: Product Effect on Complete Substitution for Smoking
Description: Number of subjects using only the assigned study product at week 6
Time Frame: 6 week post smoking substitution
Measure: Number; unit: participants
Arm/Group | Nicotine Gum | Snus
Number analyzed (Participants) | 153 | 149
participants | 56 | 56

2. Primary Outcome: Number of Cigarettes Smoked
Description: Cigarettes per day at mid intervention
Time Frame: 6 weeks post cigarette substitution
Measure: Mean (Standard Deviation); unit: cigarettes per day
Arm/Group | Nicotine Gum | Snus
Number analyzed (Participants) | 149 | 154
cigarettes per day | 18.6 (33.8) | 18.8 (28.5)

3. Primary Outcome: Number of Products Used
Description: Pieces of product per week at mid intervention
Time Frame: 6 weeks post smoking substitution
Measure: Mean (Standard Deviation); unit: Pieces per week
Arm/Group | Nicotine Gum | Snus
Number analyzed (Participants) | 149 | 154
Pieces per week | 37.6 (26.3) | 39.1 (24.0)

4. Secondary Outcome: Products Effect on Withdrawal Symptoms.
Description: Total withdrawal score on the Minnesota Nicotine Withdrawal Scale for subjects using only their assigned study product. This scale measures withdrawal symptoms from cigarettes. There are 8 items on the scale with scores that range from 0 to 4. Total score is calculated by summing the scores (excluding the craving item). Minimum score is 0 and maximum is 28. The higher the score the more severe the withdrawal.
Time Frame: Week 1-12 post switching
Population: Using assigned product only. The numbers of subjects that were only using the assigned product were 40 and 37 for nicotine gum and oral tobacco respectively at week 12. Analysis was conducted from weeks 1-12 post-switching.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Nicotine Gum | Snus
Number analyzed (Participants) | 40 | 37
units on a scale
  Baseline Scores | 4.17 (5.01) | 5.01 (5.14)
  Week 12 Scores | 5.57 (6.05) | 5.73 (6.24)

5. Secondary Outcome: Product Effect on Biomarkers of Exposure and Toxicity
Description: Total NNAL (e.g., 4-(methylnitrosamino)-1-(3-pyridyl)-1-butanol and its glucuronides) among those subjects who reported use of assigned product only (baseline and week 4 samples).
Time Frame: Baseline and Week 4 post smoking substitution
Measure: Mean (Standard Deviation); unit: pmol//mg creatinine
Arm/Group | Nicotine Gum | Snus
Number analyzed (Participants) | 58 | 52
pmol//mg creatinine
  Baseline | 1.39 (1.04) | 1.28 (0.94)
  Week 4 | 0.30 (0.39) | 1.34 (1.55)

ADVERSE EVENTS:
Time Frame: Subjects were provided study product for 12 weeks.
Arm/Group | Nicotine Gum | Snus
Serious Adverse Events (participants affected / at risk) | 1/195 | 1/196
Other Adverse Events (participants affected / at risk) | 0/195 | 0/196
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nicotine Gum (N=195) | Snus (N=196)
Death (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Subject was diagnosed with leiomyosarcoma at week 6 in the study.
Hospitalization (Psychiatric disorders) | 0 (0) | 1 (1) — Hospitalization due to suicidal ideation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes